CLINICAL TRIAL: NCT05864300
Title: Impact of Neurochecks on Sleep in Critically Ill Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jamie Labuzetta, Clinical Professor of Neurosciences, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UCSD IRB: #806351
Record Dates: First submitted 2023-05-01; First posted 2023-05-18 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Aneurysm
Keywords: neurocheck; sleep; neurological examination
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hourly Neurochecks (Active Comparator): Patients awakened for neurological exams every hour
  Interventions: Behavioral: Neurocheck frequency
- Every-Other-Hour Neurochecks (Active Comparator): Patients awakened for neurological exams every-other-hour
  Interventions: Behavioral: Neurocheck frequency

INTERVENTIONS:
Behavioral: Neurocheck frequency — Randomized to hourly or every-other-hour examinations

SUMMARY:
Background: Following acute brain injury (ABI), patients are monitored in the intensive care unit (ICU) where providers rely on frequent neurological examinations ("neurochecks") to assess for neurodeterioration. Serial neurochecks are part of guideline recommendations, but there is equipoise between hourly (Q1) and every-other-hour (Q2) evaluation. In the ICU, care-related awakenings occur frequently, but it is unclear if differential neurocheck frequencies result in differential sleep, providing the scientific premise for this proposal.

Population: Thirty patients (N=15 per group) who have undergone elective aneurysm coiling will be enrolled. On post-operative day (POD) 0, patients will be screened and approached for informed consent if they do not meet exclusion criteria, e.g., prior intracranial injury, sleep disorders, cognitive impairment, mechanical ventilation. Patients with elective aneurysm coiling are being chosen because they require ICU level of care following their intracranial procedure, but do not have structural brain injury or ongoing sedation needs that might impact sleep measurements.

Methods: Usual care: Patients are monitored every 15-30 minutes for up to 6 hours post-procedure, then Q1 or Q2 for up to 24 hours. If these patients remain stable, they are discharged home on post-operative day (POD) 1. Proposed Intervention: Enrolled patients will be randomized to Q1 or Q2 neurochecks following the institutionally required 6 hours of stable neurological and vascular checks. Once randomized, patients will undergo placement of electroencephalogram (EEG) with video, electrooculogram, and chin lead. The video EEG will be in place for at least 8 hours to include the overnight (10PM-6AM) time period. Following completion of the recording, the signals obtained will be reviewed by a blinded polysomnographic sleep technician for sleep characteristics including quantitative assessments of wakefulness, deep (N3) sleep, REM sleep, sleep efficiency, and sleep fragmentation and arousals. On POD1, patients and their nurse will fill out the Richards-Campbell Sleep Questionnaire to rate subjective sleep quality.

ELIGIBILITY:
Inclusion Criteria:

a. Adult patients who are status post uncomplicated elective coiling of unruptured cerebral aneurysm.

Exclusion Criteria:

1. Patients with past or current intracranial injury or disease.
2. Patients with known flow-limiting pathology of carotid arteries, vertebral arteries, or intracranial arteries.
3. Incomplete resolution of aneurysm.
4. Known sleep disorders (e.g., insomnia)
5. Pregnancy.
6. Incarceration.
7. Inability to communicate in English
8. Cognitive impairment or lack of decision-making capacity.
9. Ongoing sedation.
10. Mechanical ventilation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2026-01-06 (Actual); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Sleep efficiency | Within 24 hours of enrollment
  Ratio of total sleep time compared to time in bed, reported as a percentage

SECONDARY OUTCOMES:
Wakefulness | Within 24 hour of enrollment
  Blinded quantitative assessment of time spent awake
REM Sleep | Within 24 hour of enrollment
  Blinded quantitative assessment of time spent in REM sleep
Deep Sleep | Within 24 hour of enrollment
  Blinded quantitative assessment of time spent in deep sleep
Arousals | Within 24 hour of enrollment
  Blinded quantitative assessment of number of arousals (as defined by American Academy of Sleep Medicine)
Sleep quality (subjective) | Within 24 hour of enrollment
  As measured by Richards Campbell Sleep Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Health, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided